CLINICAL TRIAL: NCT00920816
Title: AG-013736 (AXITINIB) FOR THE TREATMENT OF METASTATIC RENAL CELL CANCER
Brief Title: Axitinib (AG-013736) For the Treatment of Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A4061051; 2010-018585-23 (EudraCT Number)
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Kidney Neoplasms
Keywords: Axitinib in First & Second Line Treatment of Patients With Metastatic Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Axitinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Axitinib (AG-013736)
- B (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Axitinib (AG-013736) — axitinib will be given at a starting dose of 5 mg BID with continuous dosing
  Arms: A
Drug: Sorafenib — sorafenib will be given at a dose of 400 mg BID continuous dosing
  Arms: B

SUMMARY:
The study is designed to demonstrate that axitinib (AG-013736) is superior to sorafenib in delaying tumor progression in patients with metastatic renal cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic renal cell cancer with a component of clear cell histology.
* Evidence of measurable disease.
* Patients with mRCC must have received no prior systemic first-line therapy or must have progressive disease per RECIST (version 1.0) after one prior systemic first line regimen for metastatic disease containing sunitinib, cytokine(s), or both.

Exclusion Criteria:

* Prior treatment for metastatic renal cell cancer with more that one systemic first line therapy.
* Major surgery less that 4 weeks or radiation less than 2 weeks of starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2012-07-27 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- United States (47):
  - Advanced Medical Specialties, Miami, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Indiana University Health Central Indiana Cancer Centers, Carmel, Indiana
  - Indiana University Health Central Indiana Cancer Centers, Fishers, Indiana
  - Indiana University Health Central Indiana Cancer Centers, Greenfield, Indiana
  - Indiana University Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Missouri Cancer Associates, Columbia, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - US Oncology West Region, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - Hematology-Oncology Associates of Northern NJ, PA, Parsippany, New Jersey
  - New York Oncology Hematology, PC, Albany, New York
  - New York Oncology Hematology, PC, Latham, New York
  - New York Oncology Hematology, PC, Rexford, New York
  - New York Oncology Hematology, PC, Troy, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Penn State Milton S. Hershey Medical Center, Penn State Cancer Institute, Hershey, Pennsylvania
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology- Amarillo, Amarillo, Texas
  - Texas Oncology-Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology- Bedford, Bedford, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- Fort Worth 12th Avenue, Fort Worth, Texas
  - Texas Oncology- Southwest Fort Worth, Fort Worth, Texas
  - Investigational Products Center (lPC), Fort Worth, Texas
  - US Oncology Research and Clinical Pharmacy, Fort Worth, Texas
  - Texas Oncology - Grapevine, Grapevine, Texas
  - Cancer Care Centers of South Texas, Kerrville, Texas
  - Texas Oncology- McAllen South Second Street, McAllen, Texas
  - Texas Oncology- Midland Allison Cancer Center, Midland, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology-Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology-Weslaco, Weslaco, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Christiansburg, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Low Moor, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Wytheville, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
- Bosnia and Herzegovina (3):
  - Clinic of Oncology, Banja Luka
  - Institute of Oncology, University Hospital Center Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Clinic for Oncology, Hematology and Radiotherapy, Tuzla
- Bulgaria (2):
  - Spetsializirana Bolnitsa za Aktivno Lechenie po Onkologiya, EAD, Klinika po Himioterapiya, Sofia
  - SBALOZ D-r Marko Markov-Varna, Varna
- Chile (4):
  - Instituto Clinico Oncologico del Sur, Temuco, Cautin
  - Instituto Clinico Oncologico del Sur, Temuco, Región de la Araucanía
  - Instituto de Terapias Oncologicas Providencia, Providencia, Santiago Metropolitan
  - Private Office, Santiago
- China (20):
  - Cancer Institute and Hospital ,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Haidian District, Beijing Municipality
  - The Fuzhou General Hospital, PLA Nanjing Military Area Command, Fuzhou, Fujian
  - Urology Department, Sun Yet-Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - The Oncology Department, Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Urology Department, 1st Hospital of China Medical University, Shenyang, Liaoning
  - Xijing Hospital, The Fourth Military Medical University,Oncology Department, Xi'an, Shaanxi
  - Urology Department, Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Center for Oncology, Hangzhou, Zhejiang
  - Department of Urology,Peking University First Hospital, Beijing
  - Beijing Cancer Hospital/Department of Renal Cancer and Melanoma, Beijing
  - South-Western Hospital, 3rd Military Medical University, Chongqing
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University, Cancer Hospital, Department of Urology, Shanghai
  - Tianjin Oncology Hospital,biology treatment department, Tianjin
  - Urology Department, The Second Hospital of Tianjin Medical University, Tianjin
- India (10):
  - BIBI General Hospital and Cancer Centre,, Hyderabad, Andhra Pradesh
  - Chinmaya Mission Hospital, Bangalore, Karnataka
  - Sri Venkateshwara Hospital, Bangalore, Karnataka
  - NU Hospitals, Bangalore, Karnataka
  - Cancer Care Clinic and Hospitals, Nagpur, Maharashtra
  - Shatabdi Superspeciality Hospital, Nashik, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Shettys hospital, Bangalore
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Mexico (5):
  - Hospital General de Mexico O.D., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Centro Hemato-Oncologico Privado, Toluca, State of Mexico
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Oaxaca Site Management Organization, Oaxaca City
- Philippines (5):
  - Rm. 3227 Doctors Clinic, Annex II Bldg., National Kidney & Transplant Institute, Quezon City, Diliman
  - St. Lukes Medical Center, Quezon City, National Capital Region
  - University of the East Ramon Magsaysay Memorial Medical Center, Quezon City, National Capital Region
  - Makati Medical Center, Makati City
  - Room 805, Committee on Research Room, Manila Doctors Hospital, Manila
- Romania (3):
  - Oncomed SRL, Timișoara, JUD. Timis
  - Institutul Oncologic "Prof.Dr.I.Chiricuta" Cluj-Napoca, Cluj-Napoca
  - Institutul Oncologic ''Prof.Dr. I. Chiricuta'' Cluj Napoca, Cluj-Napoca
- Russia (6):
  - GBU RO "Ryazan Regional Clinical Oncology Dispensary", Ryazan, Russian Federation
  - FGBOU VO "Ryazan State Medical University named after academician I.P.Pavlov", Ryazan, Russian Federation
  - Moscow State Healthcare Institution Oncology Clinical Dispensary #1, Moscow
  - P.A. Herzen Moscow Oncology Research Institute,, Moscow
  - FGBOU VO "First Saint-Petersburg State Medical University n.a. I.P.Pavlov", Saint Petersburg
  - Republican Clinical Oncology Dispensary of the Ministry of Health of Bashkortostan Republic, Ufa
- GVI Oncology, Port Elizabeth, South Africa
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Ukraine (5):
  - KP Dnipropetrovska oblasna klinichna likarnia im. I.I. Mechnykova" Dnipropetrovskoi oblasnoi rady,, Dnipro
  - Komunalne nekomertsiine pidpryiemstvo Kharkivskoi oblasnoi rady Oblasnyi medychnyi klinichnyi tsentr, Kharkiv
  - DU Instytut Urolohii NAMN Ukrainy, viddil onkourolohii, KNP Kyivskyi miskyi klinichnyi onkolohichnyi, Kyiv
  - Komunalne nekomertsiine pidpryiemstvo Lvivskoi oblasnoi rady Lvivskyi onkolohichnyi rehionalnyi, Lviv
  - SI "Zaporizhzhya Medical Academy of Postgraduate Education of the Ministry of Health of Ukraine", Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Rini BI, Atkins MB, Choueiri TK, Teresi RE, Rosbrook B, Thakur M, Hutson TE. Plain language summary looking at how long side effects last after treatment with axitinib is stopped in people with advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2623-2629. doi: 10.2217/fon-2023-0233. Epub 2023 Aug 1. PMID 37526095
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Rini BI, Atkins MB, Choueiri TK, Thomaidou D, Rosbrook B, Thakur M, Hutson TE. Time to Resolution of Axitinib-Related Adverse Events After Treatment Interruption in Patients With Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2021 Oct;19(5):e306-e312. doi: 10.1016/j.clgc.2021.03.019. Epub 2021 Apr 5. PMID 33947608
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Hutson TE, Al-Shukri S, Stus VP, Lipatov ON, Shparyk Y, Bair AH, Rosbrook B, Andrews GI, Vogelzang NJ. Axitinib Versus Sorafenib in First-Line Metastatic Renal Cell Carcinoma: Overall Survival From a Randomized Phase III Trial. Clin Genitourin Cancer. 2017 Feb;15(1):72-76. doi: 10.1016/j.clgc.2016.05.008. Epub 2016 May 27. PMID 27498023
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Qin S, Bi F, Jin J, Cheng Y, Guo J, Ren X, Huang Y, Tarazi J, Tang J, Chen C, Kim S, Ye D. Axitinib versus sorafenib as a second-line therapy in Asian patients with metastatic renal cell carcinoma: results from a randomized registrational study. Onco Targets Ther. 2015 Jun 8;8:1363-73. doi: 10.2147/OTT.S83302. eCollection 2015. PMID 26089686
- [Derived] Hutson TE, Lesovoy V, Al-Shukri S, Stus VP, Lipatov ON, Bair AH, Rosbrook B, Chen C, Kim S, Vogelzang NJ. Axitinib versus sorafenib as first-line therapy in patients with metastatic renal-cell carcinoma: a randomised open-label phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1287-94. doi: 10.1016/S1470-2045(13)70465-0. Epub 2013 Oct 25. PMID 24206640
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061051&StudyName=Axitinib%20%28AG-013736%29%20For%20the%20Treatment%20of%20Metastatic%20Renal%20Cell%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-line participants included all treatment-naive participants with metastatic renal cell cancer (mRCC) from global and second-line participants included all previously-treated Asian participants with mRCC.
Pre-assignment Details: All China participants were excluded from safety analysis due to inability to obtain timely approval to use data in accordance with Human Genetic Resources Administration of China (HGRAC) regulation.
Groups:
- Axitinib (First-line Participants): Participants with no prior systemic first-line therapy received axitinib (AG-013736) tablet at a starting dose of 5 milligram (mg) orally twice daily, dose adjustment was done based on the tolerability, as per investigator's discretion. Study medication was administered in cycles of 4 weeks.
- Sorafenib (First-line Participants): Participants with no prior systemic first-line therapy received sorafenib tablet at a starting dose of 400 mg orally twice daily, dose adjustment was done based on the tolerability, as per investigator's discretion. Study medication was administered in cycles of 4 weeks.
- Axitinib (Second-line Participants): Asian participants with prior systemic first-line therapy containing sunitinib or cytokine received axitinib (AG-013736) tablet at a starting dose of 5 mg orally twice daily, dose adjustment was done based on the tolerability, as per investigator's discretion. Study medication was administered in cycles of 4 weeks.
- Sorafenib (Second-line Participants): Asian participants with prior systemic first-line therapy containing sunitinib or cytokine received sorafenib tablet at a starting dose of 400 mg orally twice daily, dose adjustment was done based on the tolerability, as per investigator's discretion. Study medication was administered in cycles of 4 weeks.
Period: Overall Study
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants) | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Started | 192 | 96 | 135 | 69
Treated | 189 | 96 | 135 | 69
Participants From China (Excluded From Safety Analysis) | 16 | 8 | 124 | 64
Completed | 0 | 0 | 0 | 0
Not Completed | 192 | 96 | 135 | 69
Not completed — Death | 116 | 63 | 8 | 3
Not completed — Participant refused continued treatment for reason other than adverse events | 11 | 5 | 1 | 0
Not completed — Global deterioration of health status | 2 | 0 | 0 | 0
Not completed — Objective progression or relapse | 6 | 2 | 0 | 0
Not completed — Other | 26 | 15 | 1 | 2
Not completed — Lost to Follow-up | 11 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Data not disclosed due to lack of HGRAC filings | 16 | 8 | 124 | 64
Not completed — Randomized but not treated | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all treatment-naive participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Groups:
- Axitinib (First-line Participants): Participants with no prior systemic first-line therapy received axitinib (AG-013736) tablet at a starting dose of 5 mg orally twice daily, dose adjustment was done based on the tolerability, as per investigator's discretion. Study medication was administered in cycles of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants) | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants) | Total
Number analyzed (Participants) | 192 | 96 | 135 | 69 | 492
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 65 years | 142 | 77 | 110 | 56 | 385
  Greater than or equal to (>=) 65 years | 50 | 19 | 25 | 13 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 22 | 41 | 20 | 141
  Male | 134 | 74 | 94 | 49 | 351

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS): First-Line Participants
Description: Time in months from randomization to first documentation of objective tumor progression or death due to any cause. PFS calculated as (first event date minus date of randomization plus 1)/30.4. Tumor progression determined from oncologic assessment data (where it meets criteria for progressive disease [PD]), or from adverse event (AE) data (where outcome was "Death"). Progression using Response Evaluation Criteria in Solid Tumors (RECIST) is >= 20 percent (%) increase in sum of longest diameter of target lesions; measurable increase in non-target lesion; appearance of new lesions.
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 107)
Population: FAS included all treatment-naive participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 192 | 96
months | 10.1 [7.2 to 12.1] | 6.5 [4.7 to 8.3]
Statistical Analysis 1: Comparison: Axitinib (First-line Participants) vs Sorafenib (First-line Participants); First-line participants: hazard ratio was stratified by eastern cooperative oncology group (ECOG) performance status (0 versus 1); Test type: Superiority or Other; Hazard Ratio (HR) = 0.767, 95% CI 2-sided [0.559 to 1.053]

2. Primary Outcome: Progression Free Survival (PFS): Second-Line Participants
Description: as for outcome 1
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 103)
Population: FAS included all previously-treated Asian participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 135 | 69
months | 6.5 [4.7 to 9.1] | 4.8 [3.0 to 6.5]
Statistical Analysis 1: Comparison: Axitinib (Second-line Participants) vs Sorafenib (Second-line Participants); Second-line participants: hazard ratio was stratified by eastern cooperative oncology group (ECOG) performance status (0 versus 1) and prior treatment (sunitinib versus cytokine-containing regimen); Test type: Superiority or Other; Hazard Ratio (HR) = 0.731, 95% CI 2-sided [0.506 to 1.058]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR): First-Line Participants
Description: Percentage of participants with OR based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 107)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 192 | 96
percentage of participants | 32.3 [25.7 to 39.4] | 14.6 [8.2 to 23.3]

4. Secondary Outcome: Percentage of Participants With Objective Response (OR): Second-Line Participants
Description: as for outcome 3
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 103)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 135 | 69
percentage of participants | 23.7 [16.8 to 31.8] | 10.1 [4.2 to 19.8]

5. Secondary Outcome: Duration of Response (DR): First-Line Participants
Description: Time in months from the first documentation of objective tumor response that is subsequently confirmed to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 107)
Population: DR was calculated for the subgroup of participants from the FAS treatment-naive population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 62 | 14
months | 14.7 [11.0 to NA] — Upper limit of CI was not estimable because participants were still responding to medication as the study was ongoing at the time of primary completion analysis and this analysis was final. | 14.3 [11.3 to NA] — Upper limit of CI was not estimable because participants were still responding to medication as the study was ongoing at the time of primary completion analysis and this analysis was final.

6. Secondary Outcome: Duration of Response (DR): Second-Line Participants
Description: as for outcome 5
Time Frame: Baseline until disease progression or death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 103)
Population: DR was calculated for the subgroup of participants from the FAS previously-treated population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 32 | 7
months | NA [12.5 to NA] — Median and upper limit of CI was not estimable because participants were still responding to medication as the study was ongoing at the time of primary completion analysis and this analysis was final. | 8.7 [4.1 to NA] — Upper limit of CI was not estimable because participants were still responding to medication as the study was ongoing at the time of primary completion analysis and this analysis was final.

7. Secondary Outcome: Overall Survival (OS): First-Line Participants
Description: Time in months from date of randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 107)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 192 | 96
months | NA [18.1 to NA] — Median and upper limit of CI was not reachable as data was not matured at the time of the analysis as the study was ongoing at the time of primary completion analysis and this analysis was final. | NA [18.1 to NA] — Median and upper limit of CI was not reachable as data was not matured at the time of the analysis as the study was ongoing at the time of primary completion analysis and this analysis was final.

8. Secondary Outcome: Overall Survival (OS): Second-Line Participants
Description: as for outcome 7
Time Frame: Baseline until death (assessed on Week 6, Week 12 and thereafter every 8 weeks up to Week 103)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 135 | 69
months | 17.2 [14.8 to NA] — Upper limit of the CI was not reachable as data was not matured at the time of the analysis as the study was ongoing at the time of primary completion analysis and this analysis was final. | 18.1 [12.1 to NA] — Upper limit of the CI was not reachable as data was not matured at the time of the analysis as the study was ongoing at the time of primary completion analysis and this analysis was final.

9. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-15 (FKSI-15): First-Line Participants
Description: FKSI-15 questionnaires (lack of energy, side effects, pain, weight loss, bone pain, fatigue, enjoying life, short of breath, worsened condition, appetite, coughing, bothered by fevers, ability to work, hematuria, sleep) was used to assess quality of life (QoL) for those diagnosed with renal cell cancer. Questions answered on 5-point Likert scale: 0 to 4 (0= not at all, 1= little bit, 2= somewhat, 3= quite a bit, 4= very much). Total FKSI score 0 to 60; higher scores=better health states (Individual questions may be reversed coded, as appropriate).
Time Frame: Baseline (Pre-dose on Cycle [C]1 Day [D]1), D1 of each cycle until C23, end of treatment (up to Week 107), follow-up (28 days after last dose)
Population: FAS treatment-naive population. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants evaluated for this measure at specific time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 183 | 95
units on a scale
  C1 D1 | 43.869 (8.117) | 43.865 (6.723)
  C2 D1: number analyzed (Participants) | 176 | 90
  C2 D1 | 43.328 (7.630) | 43.969 (6.286)
  C3 D1: number analyzed (Participants) | 164 | 84
  C3 D1 | 43.366 (7.192) | 43.345 (6.878)
  C4 D1: number analyzed (Participants) | 156 | 81
  C4 D1 | 42.932 (7.566) | 42.926 (7.324)
  C5 D1: number analyzed (Participants) | 153 | 77
  C5 D1 | 43.211 (7.578) | 44.022 (6.714)
  C6 D1: number analyzed (Participants) | 141 | 72
  C6 D1 | 42.787 (8.098) | 42.344 (6.685)
  C7 D1: number analyzed (Participants) | 139 | 65
  C7 D1 | 42.474 (7.926) | 43.446 (6.931)
  C8 D1: number analyzed (Participants) | 131 | 60
  C8 D1 | 42.534 (7.510) | 44.077 (6.986)
  C9 D1: number analyzed (Participants) | 126 | 59
  C9 D1 | 42.778 (8.229) | 44.051 (7.234)
  C10 D1: number analyzed (Participants) | 122 | 55
  C10 D1 | 43.120 (7.966) | 44.018 (6.751)
  C11 D1: number analyzed (Participants) | 114 | 48
  C11 D1 | 43.264 (7.837) | 45.000 (6.130)
  C12 D1: number analyzed (Participants) | 105 | 44
  C12 D1 | 43.962 (7.243) | 45.318 (6.440)
  C13 D1: number analyzed (Participants) | 99 | 44
  C13 D1 | 44.141 (7.289) | 45.787 (6.526)
  C14 D1: number analyzed (Participants) | 95 | 37
  C14 D1 | 43.789 (7.985) | 45.459 (6.535)
  C15 D1: number analyzed (Participants) | 85 | 37
  C15 D1 | 44.176 (8.055) | 45.514 (5.914)
  C16 D1: number analyzed (Participants) | 82 | 33
  C16 D1 | 44.232 (7.515) | 46.000 (5.651)
  C17 D1: number analyzed (Participants) | 78 | 30
  C17 D1 | 43.897 (8.456) | 46.400 (6.262)
  C18 D1: number analyzed (Participants) | 71 | 28
  C18 D1 | 43.761 (8.019) | 45.357 (6.983)
  C19 D1: number analyzed (Participants) | 57 | 24
  C19 D1 | 43.737 (7.413) | 45.583 (7.366)
  C20 D1: number analyzed (Participants) | 45 | 21
  C20 D1 | 43.733 (7.605) | 44.333 (7.066)
  C21 D1: number analyzed (Participants) | 36 | 18
  C21 D1 | 45.417 (6.240) | 43.500 (7.687)
  C22 D1: number analyzed (Participants) | 23 | 12
  C22 D1 | 47.000 (5.985) | 45.833 (5.937)
  C23 D1: number analyzed (Participants) | 14 | 7
  C23 D1 | 47.571 (6.357) | 45.714 (6.651)
  End of treatment: number analyzed (Participants) | 72 | 42
  End of treatment | 39.052 (9.109) | 39.524 (8.896)
  Follow-up: number analyzed (Participants) | 41 | 26
  Follow-up | 39.683 (11.132) | 40.038 (9.897)

10. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-15 (FKSI-15): Second-Line Participants
Description: as for outcome 9
Time Frame: Baseline (Pre-dose on Cycle [C]1 Day [D]1), D1 of each cycle until C21, end of treatment (up to Week 103), follow-up (28 days after last dose)
Population: FAS previously-treated Asian population. Here 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants evaluated for this measure at specific time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 134 | 69
units on a scale
  C1 D1 | 46.753 (6.692) | 47.470 (7.450)
  C2 D1: number analyzed (Participants) | 127 | 66
  C2 D1 | 46.217 (7.028) | 45.045 (7.478)
  C3 D1: number analyzed (Participants) | 124 | 57
  C3 D1 | 45.968 (7.237) | 45.684 (7.756)
  C4 D1: number analyzed (Participants) | 116 | 53
  C4 D1 | 45.060 (8.040) | 45.792 (7.762)
  C5 D1: number analyzed (Participants) | 111 | 48
  C5 D1 | 45.775 (7.797) | 46.125 (7.491)
  C6 D1: number analyzed (Participants) | 108 | 41
  C6 D1 | 45.407 (7.274) | 46.341 (7.213)
  C7 D1: number analyzed (Participants) | 100 | 38
  C7 D1 | 45.709 (8.263) | 45.053 (7.843)
  C8 D1: number analyzed (Participants) | 89 | 37
  C8 D1 | 45.169 (7.609) | 45.676 (9.357)
  C9 D1: number analyzed (Participants) | 82 | 33
  C9 D1 | 45.829 (7.442) | 45.970 (8.487)
  C10 D1: number analyzed (Participants) | 74 | 27
  C10 D1 | 45.608 (8.299) | 46.148 (8.156)
  C11 D1: number analyzed (Participants) | 66 | 22
  C11 D1 | 45.833 (7.599) | 47.227 (6.611)
  C12 D1: number analyzed (Participants) | 59 | 22
  C12 D1 | 45.797 (6.967) | 48.091 (6.414)
  C13 D1: number analyzed (Participants) | 55 | 20
  C13 D1 | 46.727 (7.307) | 47.600 (5.762)
  C14 D1: number analyzed (Participants) | 50 | 15
  C14 D1 | 47.740 (7.094) | 49.133 (5.235)
  C15 D1: number analyzed (Participants) | 44 | 13
  C15 D1 | 48.023 (6.297) | 49.308 (4.111)
  C16 D1: number analyzed (Participants) | 38 | 12
  C16 D1 | 48.184 (6.186) | 50.500 (3.989)
  C17 D1: number analyzed (Participants) | 33 | 10
  C17 D1 | 47.909 (6.866) | 49.000 (5.869)
  C18 D1: number analyzed (Participants) | 29 | 8
  C18 D1 | 48.138 (6.791) | 49.125 (5.139)
  C19 D1: number analyzed (Participants) | 22 | 7
  C19 D1 | 48.636 (5.206) | 48.571 (7.458)
  C20 D1: number analyzed (Participants) | 21 | 6
  C20 D1 | 48.810 (6.478) | 50.500 (4.637)
  C21 D1: number analyzed (Participants) | 16 | 6
  C21 D1 | 50.188 (5.588) | 50.000 (5.177)
  End of treatment: number analyzed (Participants) | 37 | 27
  End of treatment | 41.432 (9.188) | 42.889 (8.846)
  Follow-up: number analyzed (Participants) | 13 | 12
  Follow-up | 35.385 (7.795) | 38.583 (11.556)

11. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index -Disease Related Symptoms (FKSI-DRS): First-Line Participants
Description: FKSI-DRS: subset of FKSI which is FACT-Kidney Symptom Index questionnaire used to assess QoL for participants diagnosed with renal cell cancer. FKSI contains 15 questions and FKSI-DRS 9 questions (lack of energy, pain, losing weight, bone pain, fatigue, short of breath, coughing, bothered by fevers, hematuria) each ranging from 0 (not at all) to 4 (very much). FKSI-DRS total score 0 to 36; higher scores associated with better health states (Individual questions may be reversed coded, as appropriate).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 183 | 95
units on a scale
  C1 D1 | 28.691 (5.392) | 29.653 (4.699)
  C2 D1: number analyzed (Participants) | 176 | 90
  C2 D1 | 28.728 (4.581) | 29.963 (3.817)
  C3 D1 (: number analyzed (Participants) | 164 | 84
  C3 D1 ( | 29.171 (4.093) | 29.750 (4.095)
  C4 D1: number analyzed (Participants) | 156 | 81
  C4 D1 | 28.577 (4.305) | 29.642 (4.244)
  C5 D1: number analyzed (Participants) | 153 | 77
  C5 D1 | 29.020 (4.257) | 30.255 (3.668)
  C6 D1: number analyzed (Participants) | 141 | 72
  C6 D1 | 28.574 (4.674) | 29.153 (4.009)
  C7 D1: number analyzed (Participants) | 139 | 65
  C7 D1 | 28.568 (4.548) | 29.523 (4.051)
  C8 D1: number analyzed (Participants) | 131 | 60
  C8 D1 | 28.557 (4.308) | 30.296 (3.890)
  C9 D1: number analyzed (Participants) | 126 | 59
  C9 D1 | 28.817 (4.665) | 30.186 (4.392)
  C10 D1: number analyzed (Participants) | 122 | 55
  C10 D1 | 29.057 (4.484) | 30.364 (4.143)
  C11 D1: number analyzed (Participants) | 114 | 48
  C11 D1 | 29.146 (4.207) | 30.688 (3.926)
  C12 D1: number analyzed (Participants) | 105 | 44
  C12 D1 | 29.648 (3.752) | 30.727 (3.896)
  C13 D1: number analyzed (Participants) | 99 | 44
  C13 D1 | 29.545 (4.056) | 31.483 (3.602)
  C14 D1: number analyzed (Participants) | 95 | 37
  C14 D1 | 29.579 (4.186) | 31.027 (3.790)
  C15 D1: number analyzed (Participants) | 85 | 37
  C15 D1 | 29.859 (4.438) | 30.730 (3.724)
  C16 D1: number analyzed (Participants) | 82 | 33
  C16 D1 | 29.683 (4.242) | 31.515 (3.242)
  C17 D1: number analyzed (Participants) | 78 | 30
  C17 D1 | 29.564 (4.695) | 31.567 (3.884)
  C18 D1: number analyzed (Participants) | 71 | 28
  C18 D1 | 29.380 (4.752) | 31.107 (4.425)
  C19 D1: number analyzed (Participants) | 57 | 24
  C19 D1 | 29.737 (4.414) | 31.417 (3.911)
  C20 D1: number analyzed (Participants) | 45 | 21
  C20 D1 | 29.844 (4.527) | 30.762 (4.122)
  C21 D1: number analyzed (Participants) | 36 | 18
  C21 D1 | 30.889 (3.115) | 30.056 (4.372)
  C22 D1: number analyzed (Participants) | 23 | 12
  C22 D1 | 31.696 (3.081) | 31.000 (3.275)
  C23 D1: number analyzed (Participants) | 14 | 7
  C23 D1 | 31.357 (3.388) | 31.143 (4.413)
  End of treatment: number analyzed (Participants) | 72 | 42
  End of treatment | 26.556 (5.487) | 26.786 (5.982)
  Follow-up: number analyzed (Participants) | 41 | 26
  Follow-up | 26.805 (6.373) | 26.769 (6.095)

12. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index -Disease Related Symptoms (FKSI-DRS): Second-Line Participants
Description: as for outcome 11
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 134 | 69
units on a scale
  C1 D1 | 31.020 (3.986) | 31.489 (4.538)
  C2 D1: number analyzed (Participants) | 127 | 66
  C2 D1 | 30.600 (3.892) | 30.682 (3.895)
  C3 D1: number analyzed (Participants) | 124 | 57
  C3 D1 | 30.645 (3.681) | 30.965 (3.803)
  C4 D1: number analyzed (Participants) | 116 | 53
  C4 D1 | 30.103 (4.558) | 30.679 (3.980)
  C5 D1: number analyzed (Participants) | 111 | 48
  C5 D1 | 30.676 (4.271) | 31.063 (3.629)
  C6 D1: number analyzed (Participants) | 108 | 41
  C6 D1 | 30.731 (3.973) | 31.439 (4.249)
  C7 D1: number analyzed (Participants) | 100 | 38
  C7 D1 | 30.920 (4.373) | 30.632 (4.365)
  C8 D1: number analyzed (Participants) | 89 | 37
  C8 D1 | 30.966 (4.144) | 30.703 (5.195)
  C9 D1: number analyzed (Participants) | 82 | 33
  C9 D1 | 31.012 (3.783) | 30.667 (4.884)
  C10 D1: number analyzed (Participants) | 74 | 27
  C10 D1 | 30.986 (4.133) | 30.926 (4.215)
  C11 D1: number analyzed (Participants) | 66 | 22
  C11 D1 | 31.212 (4.033) | 32.045 (3.579)
  C12 D1: number analyzed (Participants) | 59 | 22
  C12 D1 | 31.356 (3.443) | 32.000 (3.338)
  C13 D1: number analyzed (Participants) | 55 | 20
  C13 D1 | 31.418 (3.775) | 32.100 (2.989)
  C14 D1: number analyzed (Participants) | 50 | 15
  C14 D1 | 32.100 (3.321) | 32.800 (2.274)
  C15 D1: number analyzed (Participants) | 44 | 13
  C15 D1 | 32.000 (2.861) | 32.769 (2.279)
  C16 D1: number analyzed (Participants) | 38 | 12
  C16 D1 | 31.921 (3.372) | 33.167 (2.167)
  C17 D1: number analyzed (Participants) | 33 | 10
  C17 D1 | 32.061 (3.344) | 32.800 (2.898)
  C18 D1: number analyzed (Participants) | 29 | 8
  C18 D1 | 31.931 (3.116) | 32.625 (2.615)
  C19 D1: number analyzed (Participants) | 22 | 7
  C19 D1 | 32.364 (2.341) | 32.429 (4.429)
  C20 D1: number analyzed (Participants) | 21 | 6
  C20 D1 | 31.905 (2.998) | 33.500 (2.168)
  C21 D1: number analyzed (Participants) | 16 | 6
  C21 D1 | 33.125 (2.473) | 33.500 (2.345)
  End of treatment: number analyzed (Participants) | 37 | 27
  End of treatment | 28.216 (5.662) | 29.519 (4.661)
  Follow-up: number analyzed (Participants) | 13 | 12
  Follow-up | 24.692 (4.366) | 27.500 (6.762)

13. Other Pre Specified Outcome: Euro Quality of Life Questionnaire- 5 Dimensions (EQ-5D) Index Score: First-Line Participants
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 183 | 94
units on a scale
  C1 D1 | 0.710 (0.254) | 0.712 (0.272)
  C2 D1: number analyzed (Participants) | 175 | 90
  C2 D1 | 0.709 (0.214) | 0.693 (0.237)
  C3 D1: number analyzed (Participants) | 163 | 84
  C3 D1 | 0.694 (0.251) | 0.687 (0.261)
  C4 D1: number analyzed (Participants) | 156 | 81
  C4 D1 | 0.696 (0.235) | 0.668 (0.265)
  C5 D1: number analyzed (Participants) | 153 | 77
  C5 D1 | 0.708 (0.221) | 0.673 (0.269)
  C6 D1: number analyzed (Participants) | 140 | 72
  C6 D1 | 0.683 (0.263) | 0.641 (0.281)
  C7 D1: number analyzed (Participants) | 139 | 65
  C7 D1 | 0.685 (0.225) | 0.676 (0.255)
  C8 D1: number analyzed (Participants) | 131 | 60
  C8 D1 | 0.678 (0.274) | 0.717 (0.244)
  C9 D1: number analyzed (Participants) | 126 | 59
  C9 D1 | 0.704 (0.239) | 0.729 (0.202)
  C10 D1: number analyzed (Participants) | 122 | 55
  C10 D1 | 0.682 (0.277) | 0.723 (0.238)
  C11 D1: number analyzed (Participants) | 114 | 48
  C11 D1 | 0.698 (0.260) | 0.748 (0.199)
  C12 D1: number analyzed (Participants) | 105 | 44
  C12 D1 | 0.708 (0.227) | 0.742 (0.218)
  C13 D1: number analyzed (Participants) | 99 | 44
  C13 D1 | 0.708 (0.253) | 0.761 (0.220)
  C14 D1: number analyzed (Participants) | 95 | 37
  C14 D1 | 0.703 (0.260) | 0.731 (0.254)
  C15 D1: number analyzed (Participants) | 85 | 37
  C15 D1 | 0.689 (0.269) | 0.755 (0.225)
  C16 D1: number analyzed (Participants) | 82 | 33
  C16 D1 | 0.702 (0.244) | 0.775 (0.186)
  C17 D1: number analyzed (Participants) | 78 | 30
  C17 D1 | 0.706 (0.250) | 0.738 (0.250)
  C18 D1: number analyzed (Participants) | 71 | 28
  C18 D1 | 0.699 (0.259) | 0.777 (0.191)
  C19 D1: number analyzed (Participants) | 56 | 24
  C19 D1 | 0.713 (0.256) | 0.762 (0.261)
  C20 D1: number analyzed (Participants) | 45 | 21
  C20 D1 | 0.699 (0.261) | 0.710 (0.300)
  C21 D1: number analyzed (Participants) | 36 | 18
  C21 D1 | 0.712 (0.232) | 0.702 (0.307)
  C22 D1: number analyzed (Participants) | 23 | 12
  C22 D1 | 0.737 (0.255) | 0.774 (0.177)
  C23 D1: number analyzed (Participants) | 14 | 7
  C23 D1 | 0.736 (0.275) | 0.789 (0.187)
  End of treatment: number analyzed (Participants) | 70 | 42
  End of treatment | 0.635 (0.268) | 0.588 (0.291)
  Follow-up: number analyzed (Participants) | 41 | 26
  Follow-up | 0.545 (0.434) | 0.618 (0.254)

14. Other Pre Specified Outcome: Euro Quality of Life Questionnaire- 5 Dimensions (EQ-5D) Index Score: Second-Line Participants
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 134 | 69
units on a scale
  C1 D1 | 0.812 (0.225) | 0.831 (0.186)
  C2 D1: number analyzed (Participants) | 127 | 65
  C2 D1 | 0.769 (0.218) | 0.754 (0.251)
  C3 D1: number analyzed (Participants) | 124 | 58
  C3 D1 | 0.772 (0.206) | 0.755 (0.278)
  C4 D1: number analyzed (Participants) | 116 | 53
  C4 D1 | 0.737 (0.272) | 0.759 (0.211)
  C5 D1: number analyzed (Participants) | 111 | 48
  C5 D1 | 0.780 (0.203) | 0.768 (0.275)
  C6 D1: number analyzed (Participants) | 108 | 41
  C6 D1 | 0.767 (0.251) | 0.753 (0.245)
  C7 D1: number analyzed (Participants) | 100 | 38
  C7 D1 | 0.762 (0.252) | 0.768 (0.239)
  C8 D1: number analyzed (Participants) | 89 | 37
  C8 D1 | 0.758 (0.241) | 0.733 (0.339)
  C9 D1: number analyzed (Participants) | 82 | 33
  C9 D1 | 0.796 (0.203) | 0.794 (0.262)
  C10 D1: number analyzed (Participants) | 74 | 27
  C10 D1 | 0.768 (0.243) | 0.820 (0.169)
  C11 D1: number analyzed (Participants) | 66 | 22
  C11 D1 | 0.792 (0.210) | 0.848 (0.158)
  C12 D1: number analyzed (Participants) | 59 | 22
  C12 D1 | 0.797 (0.201) | 0.837 (0.157)
  C13 D1: number analyzed (Participants) | 55 | 20
  C13 D1 | 0.786 (0.217) | 0.814 (0.156)
  C14 D1: number analyzed (Participants) | 50 | 15
  C14 D1 | 0.833 (0.162) | 0.871 (0.131)
  C15 D1: number analyzed (Participants) | 44 | 13
  C15 D1 | 0.819 (0.151) | 0.829 (0.152)
  C16 D1: number analyzed (Participants) | 38 | 12
  C16 D1 | 0.811 (0.186) | 0.828 (0.142)
  C17 D1: number analyzed (Participants) | 33 | 10
  C17 D1 | 0.834 (0.158) | 0.865 (0.122)
  C18 D1: number analyzed (Participants) | 29 | 8
  C18 D1 | 0.830 (0.164) | 0.829 (0.160)
  C19 D1: number analyzed (Participants) | 22 | 7
  C19 D1 | 0.830 (0.148) | 0.861 (0.139)
  C20 D1: number analyzed (Participants) | 21 | 6
  C20 D1 | 0.832 (0.163) | 0.923 (0.129)
  C21 D1: number analyzed (Participants) | 16 | 6
  C21 D1 | 0.859 (0.155) | 0.852 (0.176)
  End of treatment: number analyzed (Participants) | 37 | 27
  End of treatment | 0.582 (0.406) | 0.623 (0.296)
  Follow-up: number analyzed (Participants) | 13 | 12
  Follow-up | 0.429 (0.358) | 0.418 (0.565)

15. Other Pre Specified Outcome: Euro Quality of Life Questionnaire- 5 Dimensions (EQ-5D) Visual Analog Scale (VAS): First-Line Participants
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0: worst imaginable health state to 100: best imaginable health state; higher scores indicate a better health state.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants)
Number analyzed (Participants) | 182 | 94
units on a scale
  C1 D1 | 71.181 (19.641) | 72.362 (16.466)
  C2 D1: number analyzed (Participants) | 175 | 90
  C2 D1 | 71.714 (16.583) | 72.422 (14.576)
  C3 D1: number analyzed (Participants) | 165 | 83
  C3 D1 | 72.006 (16.971) | 71.241 (16.252)
  C4 D1: number analyzed (Participants) | 156 | 81
  C4 D1 | 72.179 (16.980) | 72.086 (14.904)
  C5 D1: number analyzed (Participants) | 153 | 78
  C5 D1 | 72.451 (18.237) | 73.615 (14.665)
  C6 D1: number analyzed (Participants) | 141 | 72
  C6 D1 | 71.574 (18.929) | 69.944 (17.535)
  C7 D1: number analyzed (Participants) | 139 | 65
  C7 D1 | 71.050 (18.967) | 73.923 (13.998)
  C8 D1: number analyzed (Participants) | 131 | 60
  C8 D1 | 71.031 (19.081) | 73.183 (16.674)
  C9 D1: number analyzed (Participants) | 126 | 59
  C9 D1 | 72.690 (18.789) | 73.780 (16.180)
  C10 D1: number analyzed (Participants) | 122 | 55
  C10 D1 | 72.910 (19.354) | 72.400 (18.814)
  C11 D1: number analyzed (Participants) | 114 | 48
  C11 D1 | 72.763 (18.174) | 72.271 (18.512)
  C12 D1: number analyzed (Participants) | 105 | 44
  C12 D1 | 73.610 (18.275) | 75.295 (17.052)
  C13 D1: number analyzed (Participants) | 99 | 44
  C13 D1 | 73.030 (18.348) | 75.432 (17.907)
  C14 D1: number analyzed (Participants) | 95 | 37
  C14 D1 | 73.147 (17.546) | 75.108 (18.371)
  C15 D1: number analyzed (Participants) | 85 | 37
  C15 D1 | 74.494 (17.938) | 74.405 (17.650)
  C16 D1: number analyzed (Participants) | 82 | 33
  C16 D1 | 73.878 (18.289) | 75.818 (17.716)
  C17 D1: number analyzed (Participants) | 78 | 30
  C17 D1 | 73.090 (17.717) | 74.333 (18.654)
  C18 D1: number analyzed (Participants) | 71 | 28
  C18 D1 | 73.817 (17.288) | 75.571 (18.550)
  C19 D1: number analyzed (Participants) | 56 | 24
  C19 D1 | 72.089 (18.169) | 75.125 (20.919)
  C20 D1: number analyzed (Participants) | 45 | 21
  C20 D1 | 74.244 (17.044) | 74.190 (20.425)
  C21 D1: number analyzed (Participants) | 36 | 18
  C21 D1 | 75.694 (11.918) | 70.500 (21.637)
  C22 D1: number analyzed (Participants) | 23 | 12
  C22 D1 | 78.000 (12.544) | 73.917 (15.900)
  C23 D1: number analyzed (Participants) | 14 | 7
  C23 D1 | 77.143 (12.697) | 72.571 (14.820)
  End of treatment: number analyzed (Participants) | 71 | 42
  End of treatment | 67.254 (19.495) | 67.048 (22.570)
  Follow-up: number analyzed (Participants) | 41 | 26
  Follow-up | 69.195 (20.366) | 64.885 (19.916)

16. Other Pre Specified Outcome: Euro Quality of Life Questionnaire- 5 Dimensions (EQ-5D) Visual Analog Scale (VAS): Second-Line Participants
Description: as for outcome 15
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
Number analyzed (Participants) | 134 | 69
units on a scale
  C1 D1 | 82.799 (13.351) | 82.058 (14.021)
  C2 D1: number analyzed (Participants) | 127 | 65
  C2 D1 | 81.102 (13.895) | 78.231 (15.823)
  C3 D1: number analyzed (Participants) | 124 | 58
  C3 D1 | 80.895 (13.387) | 80.534 (16.453)
  C4 D1: number analyzed (Participants) | 116 | 53
  C4 D1 | 81.138 (13.508) | 81.245 (14.590)
  C5 D1: number analyzed (Participants) | 111 | 48
  C5 D1 | 83.018 (12.829) | 80.250 (15.495)
  C6 D1: number analyzed (Participants) | 108 | 41
  C6 D1 | 82.222 (13.793) | 80.829 (15.091)
  C7 D1: number analyzed (Participants) | 100 | 38
  C7 D1 | 82.900 (13.287) | 80.868 (16.140)
  C8 D1: number analyzed (Participants) | 89 | 37
  C8 D1 | 83.382 (12.636) | 81.000 (14.606)
  C9 D1: number analyzed (Participants) | 82 | 33
  C9 D1 | 84.171 (11.260) | 83.788 (10.349)
  C10 D1: number analyzed (Participants) | 74 | 27
  C10 D1 | 83.041 (13.042) | 82.778 (11.440)
  C11 D1: number analyzed (Participants) | 66 | 22
  C11 D1 | 84.136 (14.231) | 83.000 (11.832)
  C12 D1: number analyzed (Participants) | 59 | 22
  C12 D1 | 84.305 (13.211) | 83.500 (12.188)
  C13 D1: number analyzed (Participants) | 55 | 20
  C13 D1 | 82.927 (17.317) | 83.300 (11.263)
  C14 D1: number analyzed (Participants) | 50 | 15
  C14 D1 | 86.520 (10.831) | 86.667 (8.715)
  C15 D1: number analyzed (Participants) | 44 | 13
  C15 D1 | 85.841 (11.783) | 86.462 (8.678)
  C16 D1: number analyzed (Participants) | 38 | 12
  C16 D1 | 87.579 (10.391) | 86.083 (8.816)
  C17 D1: number analyzed (Participants) | 33 | 10
  C17 D1 | 88.424 (10.866) | 84.300 (10.328)
  C18 D1: number analyzed (Participants) | 29 | 8
  C18 D1 | 86.586 (13.605) | 83.125 (8.839)
  C19 D1: number analyzed (Participants) | 22 | 7
  C19 D1 | 89.500 (8.684) | 82.143 (11.495)
  C20 D1: number analyzed (Participants) | 21 | 6
  C20 D1 | 90.333 (8.679) | 86.000 (9.695)
  C21 D1: number analyzed (Participants) | 16 | 6
  C21 D1 | 90.313 (9.741) | 84.167 (9.704)
  End of treatment: number analyzed (Participants) | 37 | 27
  End of treatment | 75.568 (17.934) | 74.741 (17.623)
  Follow-up: number analyzed (Participants) | 13 | 12
  Follow-up | 58.154 (20.760) | 64.333 (25.564)

ADVERSE EVENTS:
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety is reported for all participants excluding participants from China, who received at least 1 dose of study drug with treatment assignments designated according to actual study drug received.
Arm/Group | Axitinib (First-line Participants) | Sorafenib (First-line Participants) | Axitinib (Second-line Participants) | Sorafenib (Second-line Participants)
All-Cause Mortality (participants affected / at risk) | 117/173 | 63/88 | 9/11 | 3/5
Serious Adverse Events (participants affected / at risk) | 77/173 | 26/88 | 6/11 | 3/5
Other Adverse Events (participants affected / at risk) | 161/173 | 83/88 | 11/11 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (First-line Participants) (N=173) | Sorafenib (First-line Participants) (N=88) | Axitinib (Second-line Participants) (N=11) | Sorafenib (Second-line Participants) (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Disease progression (General disorders) | 20 | 6 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Axonal and demyelinating polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (First-line Participants) (N=173) | Sorafenib (First-line Participants) (N=88) | Axitinib (Second-line Participants) (N=11) | Sorafenib (Second-line Participants) (N=5)
Hypothyroidism (Endocrine disorders) | 36 | 5 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 8 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 32 | 7 | 2 | 0
Constipation (Gastrointestinal disorders) | 17 | 10 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 88 | 34 | 6 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 38 | 15 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 20 | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 38 | 11 | 0 | 0
Chest pain (General disorders) | 9 | 7 | 1 | 1
Fatigue (General disorders) | 55 | 25 | 4 | 2
Pyrexia (General disorders) | 9 | 4 | 2 | 0
Nasopharyngitis (Infections and infestations) | 10 | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 19 | 8 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 17 | 8 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 6 | 0 | 0
Blood creatinine increased (Investigations) | 14 | 6 | 2 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 17 | 2 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 70 | 24 | 4 | 1
Lipase increased (Investigations) | 7 | 5 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 48 | 16 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 10 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 14 | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 6 | 4 | 0
Proteinuria (Renal and urinary disorders) | 19 | 9 | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 14 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 37 | 10 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 11 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 17 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 41 | 31 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 15 | 18 | 1 | 0
Hypertension (Vascular disorders) | 83 | 28 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 15 | 9 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 9 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 10 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 13 | 3 | 1 | 0
Asthenia (General disorders) | 41 | 15 | 5 | 0
Mucosal inflammation (General disorders) | 21 | 9 | 1 | 0
Oedema peripheral (General disorders) | 10 | 4 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 3 | 1
Dizziness (Nervous system disorders) | 14 | 2 | 1 | 0
Headache (Nervous system disorders) | 23 | 6 | 1 | 0
Anxiety (Psychiatric disorders) | 10 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 10 | 5 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 21 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 6 | 1 | 0
Hypotension (Vascular disorders) | 13 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 5 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 10 | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 10 | 4 | 2 | 0
Haemorrhoid infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood calcium increased (Investigations) | 0 | 0 | 1 | 0
Blood chloride increased (Investigations) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 2 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0
Haematocrit increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1 | 2
Lymphocyte percentage decreased (Investigations) | 0 | 0 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 1 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Anisocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Polychromasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dizziness exertional (Nervous system disorders) | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 10 | 0 | 1 | 0
Mucosal excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Haemostasis (Surgical and medical procedures) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The objective of the statistical analysis for secondary endpoints was to summarize data using descriptive statistics without performing any hypothesis testing. Safety analysis did not include data from all China participants due to inability to obtain timely approval to use data in accordance to HGRAC regulations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.